CLINICAL TRIAL: NCT06516094
Title: Efficacy and Safety Study of Celecoxib / Pregabalin / Vitamin B Fixed Dose Combination Versus Celecoxib + Vitamin B Versus Pregabalin + Vitamin B in the Management of Chronic Low Back Pain Mixed Component
Brief Title: Efficacy and Safety in the Combination of Celecoxib / Pregabalin / Vitamin B for Low Back Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30222-III-22 (1)
Record Dates: First submitted 2024-06-26; First posted 2024-07-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain
Keywords: Low-back pain; Chronic pain; Vitamin B; Pregabalin; Celecoxib
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Celecoxib; Folic Acid; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Celecoxib+Pregabalin+Vitamin B(thiamine mononitrate/pyridoxone hydrochloride/cyanocobalamin)+Placebo (Experimental): Administered orally, 1 tablet + 1 capsule a day, for 3 months.
  Interventions: Drug: Celecoxib+Pregabalin+Vitamin B fixed dose
- Celecoxib + Vitamin B (thiamine mononitrate/ pyridoxone hydrochloride/ cyanocobalamin) (Active Comparator): Administered orally, 1 capsule + 1 tablet a day, for 3 months
  Interventions: Drug: Celecoxib + Vitamin B fixed dose
- Pregabalin + Vitamin B (thiamine mononitrate/ pyridoxone hydrochloride/ cyanocobalamin) (Active Comparator): Administered orally, 1 capsule + 1 tablet a day, for 3 months
  Interventions: Drug: Pregabalin + Vitamin B fixed dose

INTERVENTIONS:
Drug: Celecoxib+Pregabalin+Vitamin B fixed dose — One tablet of 200 mg / 150 mg / 100 mg / 50 mg / 0.50 mg + 1 capsule of placebo once a day
  Other Names: Cele+Pre+Vit B
  Arms: Celecoxib+Pregabalin+Vitamin B(thiamine mononitrate/pyridoxone hydrochloride/cyanocobalamin)+Placebo
Drug: Celecoxib + Vitamin B fixed dose — One capsule of 200 mg + 1 tablet of 100 mg / 50 mg / 0.50 mg once a day
  Other Names: Cele+Vit B
  Arms: Celecoxib + Vitamin B (thiamine mononitrate/ pyridoxone hydrochloride/ cyanocobalamin)
Drug: Pregabalin + Vitamin B fixed dose — One capsule of 150 mg + 1 tablet of 100 mg / 50 mg / 0.50 mg once a day
  Other Names: Pre+Vit B
  Arms: Pregabalin + Vitamin B (thiamine mononitrate/ pyridoxone hydrochloride/ cyanocobalamin)

SUMMARY:
Phase III longitudinal, multicenter, randomized, double-blind clinical trial. The aim of this study is to evaluate the efficacy and security of the drug combination of Celecoxib / Pregabalin / Vitamin B versus Celecoxib + Vitamin B, versus Pregabalin + Vitamin B in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
Researchers will compare the fixed-dose combination of Celecoxib/Pregabalin/Vitamin B versus Celecoxib + Vitamin B versus Pregabalin + Vitamin B for chronic low back pain. The adverse events related to the interventions would be registered in each follow up visit.

Participants will:

* Be randomized into one of the 3 intervention groups (A,B,C) once a day for 12 weeks
* If needed the dose could be escaleted twice a day.
* Visit the clinic at weeks 2, 4, 8 and 12 for checkups and follow up

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study and give written informed consent
* Subjects must have chronic low back pain with a high probability of a significant neuropathic component during 4 years or less (but not less than 3 months)
* Patients with chronic low back pain reported as moderate to severe intensity (EVA ≥ 40 mm)
* Patients with Neuropathic Pain Questionnaire (DN4) result ≥ 4
* Women of childbearing potential under a medically acceptable method of contraception

Exclusion Criteria:

* Patients participating in another clinical trial involving an investigational treatment or participation in one within 4 weeks prior to study start
* Patients whose participation in the study may be influenced (employment relationship with the research site or sponsor, inmates, etc.)
* At medical discretion, a disease that affects prognosis and prevents outpatient management, for example, but not limited to: end-stage cancer, kidney, heart, respiratory or liver failure, mental illness or with scheduled surgical or hospital procedures
* History/presence of any disease or condition that, in the opinion of the Investigator, could pose a risk for the patient or confusing the efficacy and safety of the investigational product
* Patients in whom the study drug is contraindicated for medical reasons
* Patients with allergy or hypersensitivity to the active substance of the study drugs, related products or excipients
* Pregnant women, women breastfeeding or planning a pregnancy during the conducting the study
* Significant history of gastrointestinal diseases (e.g., gastric ulcer, Crohn's disease, Ulcerative Colitis, etc.)
* Current treatment with opioids and/or NSAIDs including COX-2 inhibitors (except celecoxib), reported in clinical history in the last 24 hours to the signing of the informed consent
* Patients who are receiving monoamineoxidase inhibitors (MAOIs) or who have received them in the course of the 2 weeks prior to signing the informed consent
* Patients with a history of alcohol or drug abuse in the last year
* Patients with a history of ischemic heart disease, peripheral artery disease, and/or cerebral vascular disease (including patients who have recently undergone coronary revascularization or angioplasty)
* Patients with a history of seizures, epileptic status and/or grand mal seizures
* History of chronic liver failure Child-Pugh A, B, and/or C
* History of acute renal failure (glomerular filtration rate <30 ml/min/1.72 m2)
* Patient with a history of chronic pain associated with fibromyalgia, Paget's disease or bone pain induced by metastatic cancer
* History of major trauma to the lower back in the past 14 days
* Low back pain due to a visceral disorder (e.g., dysmenorrhea, history of endometriosis)
* Patients with a history of orthopedic surgery of the lumbar region secondary to chronic low back pain
* Patients with symptoms suggestive of COVID-19 infection (fever, cough, dyspnea) and/or contact in the last 14 days with a suspected or positive patient for COVID-19

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage change of Celecoxib / Pregabalin / Vitamin B Combination versus Celecoxib + Vitamin B versus Pregabalin + Vitamin B in the management of chronic low back pain through the visual analog pain scale (VAS). | 3 months
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. At the end of the clinical trial the change porcentage will be measured and compared between treatment groups.
Number of participants with treatment-related adverse events through the patient's diary record. | 3 months
  To describe the frequency, intensity and causality of the adverse events presented during the clinical trial by treatment group. The adverse events will be registered by the patient in the diary record. Each adverse event will be followed up at the discretion of the researcher.

SECONDARY OUTCOMES:
To describe the sociodemographic characteristics of the patients included in the study by treatment group | 3 months
  A general description of sex, age, race, weight, height and BMI.
  * Body weight: should be obtained on a scale, with the patient without shoes, in a standing position it would be recorded in kilograms.
  * Height: must be obtained with a stadimeter, with the patient without shoes, in a standing position, the record will be in meters Height will be measured only at visit 0, and will be taken as a reference for measurement of BMI.
  * BMI: calculated with the formula: Weight/height2 and will be recorded in kg/m2.
  Weight and height will be combined to report BMI in kg/m^2
Assess the proportion of patients who reported >30% improvement in pain intensity measured through VAS at 12 weeks per treatment group | 3 months
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. At the end of the clinical trial the proportion of patiens with an improvement of pain >30% will be reported and compared between treatment groups.
Assess the proportion of patients who reported >50% improvement in pain intensity measured through VAS at 12 weeks per treatment group | 3 months
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess pain intensity. At the end of the clinical trial the proportion of patiens with an improvement of pain >50% will be reported and compared between treatment groups.
Assess at what time of follow-up the greatest reduction in pain intensity was achieved, measured through VAS, per treatment group. | 3 months
  The visual analog pain scale (VAS) is a straight line in which one end signifies absence of pain and the other means the worst pain imaginable. The researcher will apply the VAS scale to each patient at each visit to assess time of greatest reduction in pain intensity.
Assess and compare the degree of physical disability due to low back pain, measured through the Oswestry disability questionnaire at 4 and 12 weeks per treatment group. | 3 months
  The Oswestry questionnaire has been designed to give us information as to how the back pain has affected the ability to manage everyday life of patients, it classifies QOL as: no disability, mild disability, moderate disability, severe disability and completely disabled. The disability degree would be compared.
Assess and compare the degree of disability to perform daily activities due to low back pain, reported through Roland-Morris questionnaire at 4 and 12 weeks per group treatment | 3 months
  The Roland-Morris questionnaire has been designed to assess the activities of daily living functional mobility pain. A maximum score of 24 indicates the greatest degree of disability from pain. The disability degree would be compared.
Assess and compare health status through the 5-level, 5-dimensions EuroQol questionnaire (EQ-5D-5L) at 12 weeks from baseline in each group of treatment | 3 months
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS)The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'.
Report the number of patients that required dose escalation | 3 months
  Dose escalation criteria:
  1. Increase in VAS values compared to the previous visit.
  2. Use of rescue medication at least in three consecutive occasions.
  3. Percentage of adherence to treatment ≥ 80% The researcher will assess the need for dose escalation or not in each visit.
Report the number of patients who require the use of rescue medication during the clinical trial by treatment group. | 3 months
  The rescue medication will be tramadol 50 mg:
  - The patient that considers the need for rescue medication must call the doctor, who will be in charge of applying the VAS scale by telephone. If the doctor considers it necessary, the taking of the rescue medication will be indicated.
Report the number of patients who presented therapeutic failure during the study among the treatment groups | 3 months
  Therapeutic failure will be defined by the principal researcher previous medical consult, the following criteria must be present:
  * Increase in the parameters of the VAS scale at 12 weeks from baseline
  * ≥80% to adherence to treatment
  * The consumption of at least 2 doses of the designated group treatment
  * The need of use of the rescue medication during 24 consecutive hours
  * The absence of comorbidities that could increase the pain (knew traumatism during the clinical trial)
To report the percentage of therapeutic adherence at 12 weeks of intervention by group of treatment. | 3 months
  Therapeutic adherence will be defined by the principal researcher. Adherence to treatment will be defined as a consumption ≥ 80% of the doses that the patient should have ingested at the time of the corresponding evaluation.
Blood concentration of BUN of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting BUN parameters. Comparisons of serum levels between groups will be made.
Blood concentration of glucose of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting glucose parameters. Comparisons of serum levels between groups will be made.
Blood concentration of urea of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting urea parameters. Comparisons of serum levels between groups will be made.
Blood concentration of creatinin of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting creatinin parameters. Comparisons of serum levels between groups will be made.
Blood concentration of Alkaline Phosphatase of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting Alkaline Phosphatase parameters. Comparisons of serum levels between groups will be made.
Blood concentration of total bilirrubin of the patients included in the study by treatment group | 3 months
  A blood sample will be taken in each visit reporting total bilirrubin parameters. Comparisons of serum levels between groups will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Juan L Torres-Méndez, Principal Investigator — Clínica de Ozonoterapia RGH, A.C.; Raul Coca-Nuñez, Principal Investigator — CICMEX; Adelfia Urenda-Quezada, Principal Investigator — Imacen S.A. de C.V.; Ma. Dolores Alonso-Martinez, Principal Investigator — Servicios Avanzados de Investigación Medica Mediadvance S.C.; Ramon F Villalobos-Bojorquez, Principal Investigator — Clinical Research Institute, S.C.; Rodrigo Suárez-Otero, Principal Investigator — Consultorio Médico "Dr. Rodrigo Suárez Otero"
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponce-Monter HA, Ortiz MI, Garza-Hernandez AF, Monroy-Maya R, Soto-Rios M, Carrillo-Alarcon L, Reyes-Garcia G, Fernandez-Martinez E. Effect of diclofenac with B vitamins on the treatment of acute pain originated by lower-limb fracture and surgery. Pain Res Treat. 2012;2012:104782. doi: 10.1155/2012/104782. Epub 2011 Oct 31. PMID 22135737
- [Background] Antonucci R, Zaffanello M, Puxeddu E, Porcella A, Cuzzolin L, Pilloni MD, Fanos V. Use of non-steroidal anti-inflammatory drugs in pregnancy: impact on the fetus and newborn. Curr Drug Metab. 2012 May 1;13(4):474-90. doi: 10.2174/138920012800166607. PMID 22299823
- [Result] Raffaeli W, Arnaudo E. Pain as a disease: an overview. J Pain Res. 2017 Aug 21;10:2003-2008. doi: 10.2147/JPR.S138864. eCollection 2017. PMID 28860855
- [Result] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Result] Kongsted A, Kent P, Axen I, Downie AS, Dunn KM. What have we learned from ten years of trajectory research in low back pain? BMC Musculoskelet Disord. 2016 May 21;17:220. doi: 10.1186/s12891-016-1071-2. PMID 27209166
- [Result] Morlion B. Pharmacotherapy of low back pain: targeting nociceptive and neuropathic pain components. Curr Med Res Opin. 2011 Jan;27(1):11-33. doi: 10.1185/03007995.2010.534446. Epub 2010 Nov 18. PMID 21083513
- [Result] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Result] Ho KY, Gwee KA, Cheng YK, Yoon KH, Hee HT, Omar AR. Nonsteroidal anti-inflammatory drugs in chronic pain: implications of new data for clinical practice. J Pain Res. 2018 Sep 20;11:1937-1948. doi: 10.2147/JPR.S168188. eCollection 2018. PMID 30288088
- [Result] Ajmone-Cat MA, Bernardo A, Greco A, Minghetti L. Non-Steroidal Anti-Inflammatory Drugs and Brain Inflammation: Effects on Microglial Functions. Pharmaceuticals (Basel). 2010 Jun 14;3(6):1949-1965. doi: 10.3390/ph3061949. PMID 27713336
- [Result] Wishart DS, Feunang YD, Guo AC, Lo EJ, Marcu A, Grant JR, Sajed T, Johnson D, Li C, Sayeeda Z, Assempour N, Iynkkaran I, Liu Y, Maciejewski A, Gale N, Wilson A, Chin L, Cummings R, Le D, Pon A, Knox C, Wilson M. DrugBank 5.0: a major update to the DrugBank database for 2018. Nucleic Acids Res. 2018 Jan 4;46(D1):D1074-D1082. doi: 10.1093/nar/gkx1037. PMID 29126136
- [Result] Gong L, Thorn CF, Bertagnolli MM, Grosser T, Altman RB, Klein TE. Celecoxib pathways: pharmacokinetics and pharmacodynamics. Pharmacogenet Genomics. 2012 Apr;22(4):310-8. doi: 10.1097/FPC.0b013e32834f94cb. No abstract available. PMID 22336956
- See also: Low back pain — http://doi.org/10.1016/S0140-6736(21)00733-9
- See also: Non-steroidal anti-inflammatory drugs: an overview — http://doi.org/10.22270/jddt.v9i1-s.2287
- See also: Nonsteroidal anti-inflammatory drugs in chronic pain: implications of new data for clinical practice — http://doi.org/10.2147/JPR.S168188
- See also: National Center for Biotechnology Information (2022). PubChem Compound Summary for CID 2662, Celecoxib — http://pubchem.ncbi.nlm.nih.gov/compound/Celecoxib
- See also: National Center for Biotechnology Information — http://pubchem.ncbi.nlm.nih.gov/compound/Pregabalin
- See also: National Center for Biotechnology Information (2022). PubChem Compound Summary for CID 1130, Thiamine — http://pubchem.ncbi.nlm.nih.gov/compound/Thiamine
- See also: National Center for Biotechnology Information (2022). PubChem Compound Summary for CID 1054, Pyridoxine — http://pubchem.ncbi.nlm.nih.gov/compound/Pyridoxine
- See also: National Center for Biotechnology Information (2022). PubChem Compound Summary for CID 5311498, Cyanocobalamin — http://pubchem.ncbi.nlm.nih.gov/compound/Cyanocobalamin
- See also: Sample Size Calculator — http://www.gigacalculator.com/calculators/power-sample-size-calculator.php